CLINICAL TRIAL: NCT01961713
Title: Circulating Tumor Cell Analysis in Patients With Localized Prostate Cancer Undergoing Prostatectomy
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Prostate Cancer Foundation Clinical Research Consortium (Network)
Responsible Party: Principal Investigator, Richard J. Lee, MD, Assistant Physician, Massachusetts General Hospital
Other Study IDs: 08-207
Record Dates: First submitted 2010-09-30; First posted 2013-10-11 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: circulating tumor cells; CTC-Chip
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prostatectomy: Subjects with prostate cancer diagnosed on prostate biopsy who undergo radical prostatectomy at Massachusetts General Hospital

SUMMARY:
This study will evaluate a method to detect tumor cells that are circulating in the blood without getting a biopsy. The investigators already know from other studies that cancer tumors shed a small number of cells into the bloodstream every day. These are called circulating tumor cells (CTCs). Some early studies indicate the amount and type of CTCs in the blood can help determine the status of the tumor itself and the way it is responding to treatment. In this study, the investigators will compare the number of CTCs in the blood at different time frames before and after surgery to remove the prostate.

DETAILED DESCRIPTION:
The investigators will collect a blood sample for the study when the participant has other blood tests drawn for their cancer treatment. The investigators will take one sample to check prostate specific antigen (PSA) levels and another blood sample for CTC analysis. The investigators will be drawing blood at the following time points: Screening; One day after surgery; 7-14 days after surgery; 3-6 months after surgery; at PSA recurrence or at two years.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years of age or older
* Pathologically confirmed diagnosis of prostate adenocarcinoma
* Non-metastatic prostate cancer
* Planned radical prostatectomy at Massachusetts General Hospital

Exclusion Criteria:

* Patients must not have received prior radiation therapy, hormone therapy, or other medical therapy for prostate cancer prior to prostatectomy. Post-prostatectomy therapy at the discretion of the patient's treating physician(s) is allowed.
* Patients must not have metastatic prostate cancer
* No prior or current diagnosis of epithelial malignancy, except for skin cancer (squamous cell carcinoma or basal cell carcinoma)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer that will be undergoing prostatectomy at Massachusetts General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between CTC quantity and pathologic stage | Up to 2 weeks after prostatectomy
  To evaluate the relationship between pre-operative CTC quantity and pathologic stage in men with early stage prostate cancer undergoing prostatectomy. Processing of the pathology specimen will require up to 2 weeks after surgery.
Persistent CTC and biochemical recurrence | 2 year
  To examine the relationship between persistent CTCs and biochemical recurrence after radical prostatectomy for localized prostate cancer

SECONDARY OUTCOMES:
Compare chromosome translocation status | 2 years
  To compare the chromosome translocation status (TMPRSS2 fusion with ETS-related genes ERG, ETV1, ETV4, or ETV5) in CTCs with the primary tumor, and examine potential correlations between specific chromosomal translocations with biochemical recurrence.
Explore other uses of CTCs captured | 10 years
  To explore hypotheses about other uses of the CTCs captured with teh CTC-Chip, or the RNA or protein isolated from the CTCs, from the patients with localized prostate cancer for potential research and clinical applications.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Lee, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachsuetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No